CLINICAL TRIAL: NCT03036735
Title: Rates of Middle Meatus (MM) Synechiae Formation Post Endoscopic Sinus Surgery (ESS)
Brief Title: Rates of Middle Meatus Synechiae Formation Post ESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funds
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: SinuSys Corporation (Industry)
Responsible Party: Principal Investigator, Peter Catalano, Director otolaryngology, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00723
Record Dates: First submitted 2015-05-04; First posted 2017-01-30 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Intervention Model Description: Subjects undergoing endoscopic sinus surgery (ESS) will receive one steroid eluting spacer placed into the surgical site on one side, and one spacer without steroid placed on the other side.
Masking Description: At the end of surgery, the Surgery Fellow will insert either the Drug Eluting Spacer or the Silastic spacer into each side of the subject's nose. The subject will receive one of each spacer. The fellow will record which spacer was placed on which side using a special coding system to keep this information private. This maintains the blinding for the primary surgeon/outcome assessor and subject.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Steroid Eluting Spacer (Experimental): Subjects will receive one steroid eluting spacer (Restora Mometasone Furate Eluting Spacer) placed into the surgical site on one side, and one spacer without drug (Silastic spacer) placed on the other side.
  The Restora Mometasone Furate Eluting Spacer will be compared to the Silastic spacer.
  Interventions: Device: steroid eluting spacer

INTERVENTIONS:
Device: steroid eluting spacer — The Restora Mometasone Furate Eluting Spacer will be compared to the Silastic spacer.

SUMMARY:
The study is designed to evaluate if addition of the steroid to the spacer / stent will improve healing after endoscopic sinus surgery (ESS) compared to spacer without drug.

DETAILED DESCRIPTION:
The study is designed to evaluate basic device usability and confirm safety and effectiveness of the Restora Steroid Eluting spacer compared to a Silastic spacer.

At the completion of their procedure, patients undergoing ESS will receive one steroid eluting spacer placed into the surgical site on one side, and one spacer without drug placed on the other side. Patients will return for standard post-op visits. Between post-op day 6 and 8, both spacers will be removed. Patients will again be seen on post-op day 35 and 90 to evaluate the surgical sites with respect to healing, scarring, infection, degree of inflammation, polyp formation, and the need for secondary intervention. Data from the two sides will be compared to determine if there is a benefit derived from the spacer with steroid vs the one without.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Diagnosis of chronic rhinosinusitis (CRS), per current guidelines
3. Patients who need to undergo primary bilateral complete endoscopic sinus surgery
4. Subject has the ability to follow the study instructions, is willing to be available on the specific required study visit days, and is willing to complete all study visit procedures and assessments
5. Subject must understand the research nature of this study and sign an informed consent prior to the performance of any study-specific procedure or assessment

Exclusion Criteria

1. Subject is pregnant or breast feeding
2. Patients with sino-nasal tumors
3. Patients solely undergoing nasal septal reconstruction
4. Patients with previous history of endoscopic sinus surgery
5. Cystic fibrosis or syndromic patients
6. Patients with autoimmune diseases
7. Patients who have taken oral steroids less than 30 days prior to surgery
8. Patients with a history or diagnosis of glaucoma or ocular hypertension
9. Any other circumstance or condition that in the Investigator's opinion causes the subject to be an inappropriate candidate for participating in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04-05 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated prematurely
Groups:
- Drug Eluding Spacer: Restora Mometasone Furate spacer
Period: Overall Study
Arm/Group | Drug Eluding Spacer
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Groups:
- Drug Eluding Spacer: nasal drug eluding spacer
Arm/Group | Drug Eluding Spacer
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Middle Meatal Synechiae Post Fess ( Functional Endoscopic Surgery )," as Accurate and Appropriate).
Description: Steroid eluting spacer will be measured by incidence of 35 and 90-day post Functional Endoscopic Sinus Surgery (FESS) incidence of middle meatal synechiae.
Time Frame: 35 to 90days
Population: Study was terminated , funds withdrawn. No data was collected or analyzed.
Arm/Group | Drug Eluding Spacer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: study was terminated and funds with drawn. No data was obtained.
Groups:
- Steroid Eluting Spacer: Subjects will receive one steroid eluting spacer (Restora Mometasone Furate Eluting Spacer) placed into the surgical site on one side, and one spacer without drug (Silastic spacer) placed on the other side.
  The Restora Mometasone Furate Eluting Spacer will be compared to the Silastic spacer.
  steroid eluting spacer: The Restora Mometasone Furate Eluting Spacer will be compared to the Silastic spacer.
Arm/Group | Steroid Eluting Spacer
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid Eluting Spacer (N=0)
Study was terminated for lack of funds (Ear and labyrinth disorders) | 0 (0) — Study was terminated prematurely for lack of funds

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No